CLINICAL TRIAL: NCT01125670
Title: Pharmacokinetic Study of YM150 - A Pharmacokinetic Study to Investigate the Effect of Food on the Pharmacokinetics of YM150 Tablet-
Brief Title: A Pharmacokinetic Study to Investigate the Effect of Food on the Pharmacokinetics of YM150 Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 150-CL-047
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Healthy Volunteer; Pharmacokinetics of YM150
Keywords: YM150; Food effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fast-fed sequence group (Experimental)
  Interventions: Drug: YM150
- fed-fast sequence group (Experimental)
  Interventions: Drug: YM150

INTERVENTIONS:
Drug: YM150 — oral

SUMMARY:
This study is to evaluate the effect of food on the pharmacokinetics of YM150 in healthy make adult subjects.

DETAILED DESCRIPTION:
To evaluate the effect of food on the pharmacokinetics of YM150 in healthy non-elderly adult male subjects using a 2×2 crossover design. Also, to evaluate the safety of YM150.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: ≥50.0 kg, <80.0 kg
* BMI: ≥17.6, <26.4
* Healthy, as judged by the investigator or sub-investigator based on the results of physical examinations and lab tests

Exclusion Criteria:

* Received any investigational drugs within 120 days before the study
* Donated 400 mL of whole blood within 90 days, 200 mL of whole blood within 30 days, or blood components within 14 days before the study
* Received medication within 7 days before the study
* A deviation from the assessment criteria of physical examinations or laboratory tests
* A deviation from the normal reference range of coagulation test [PT (INR) or aPTT]
* History of drug allergies
* Upper gastrointestinal disease within 7 days before the study
* Concurrent or previous hepatic, gastrointestinal, heart, cerebrovascular or respiratory diseases
* Concurrent or previous malignant tumor
* Previous treatment with YM150

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of YM150 and its metabolites measured by blood samples | for 3 days after drug administration

SECONDARY OUTCOMES:
Safety assessed by AEs, vital signs, 12-lead ECG and lab tests | for 3 days after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kyushu, Japan